CLINICAL TRIAL: NCT03075917
Title: Validation of an Allergic Rhinitis Control Test in Children
Acronym: ARCTEnfants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL16_0283
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): questionnaire for allergic rhinitis control children from 5 to 11 years old who complete a self questionnaire regarding allergic rhinitis control during the consultation and after 15 days
  Interventions: Other: Self Questionnaire

INTERVENTIONS:
Other: Self Questionnaire — self questionnaire for allergic rhinitis control

SUMMARY:
Allergic rhinitis is a common condition that affects adults as well as children and adolescents, often with impaired quality of life. Patients often report a poor level of satisfaction with the effectiveness of their treatment and are always looking for more drug combinations to improve their symptom. Several tools exist for assessing control of allergic rhinitis, but none has been validated in teenagers or in children. A study conducted in 2008, resulted in the validation of a self-administered control test of allergic rhinitis (ARCT) in patients from 12 years of age. We propose to adapt ARCT adult to pediatric population from 5 to 11 years old.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 to 11 years old, consulting a practitioner for an allergic rhinitis
* Parents formulated their study participation agreement by signing the consent form.

Exclusion Criteria:

* Patients that are already treated for the actual episode of allergic rhinitis and are satisfied of the treatment.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Score of the allergic rhinitis control self questionnaire | 15 days
  Score of the allergic rhinitis control self questionnaire in teenagers from 5 to 11 years old.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH Louis Pasteur, Bagnols-sur-Cèze
  - Maison de santé de Lasalle, Lasalle
  - CH de MILLAU, Millau
  - Centre (Ctre) Medical Ravas - Malbosc, Montpellier
  - University hospital of Montpellier, Montpellier
  - Hôpital Trousseau,, Paris

IPD SHARING:
Plan to Share IPD: No